CLINICAL TRIAL: NCT02424890
Title: Trial of Multidisciplinary Team Stress and Performance in Immersive Simulation for Management of Infant in Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Sim-stress.1
Record Dates: First submitted 2015-03-19; First posted 2015-04-23 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Stress

ARMS (2):
- Repetitive Sim Group (Active Comparator): 9 simulation sessions
  Interventions: Other: MDT simulation sessions of management of life-threatening events over 1 year
- Control Group (Active Comparator): 3 simulation sessions
  Interventions: Other: MDT simulation sessions of management of life-threatening events over 1 year

INTERVENTIONS:
Other: MDT simulation sessions of management of life-threatening events over 1 year — 9 simulation sessions over 1 year for Repetitive Sim Group and 3 simulation sessions over 1 year for Control Group

SUMMARY:
The objective of this randomized trial is to study the effect of stress on performance and the effect of repetition of simulation sessions on performance and stress. This study is a randomized controlled trial including 48 participants who composed 12 multidisciplinary teams (MDTs). Each MDT was made up of 4 persons: an emergency physician, a resident, a nurse, and an ambulance driver who usually compose an emergency team of the French Emergency Medical Service (EMS). 6 MDTs underwent 9 simulation sessions over 1 year (Repetitive SIm Group). 6 MDTs underwent 3 simulation sessions over 1 year (Control Group). Evidence of the existence of stress was assessed in 3 ways: salivary cortisol, Holter parameters, and psychological stress questionnaires. The impact of stress on overall team performance, on technical procedure, and on teamwork, is evaluated by specific validated scales. Detection of post-traumatic stress (PTSD) is performed by self-evaluation on the 7th day and after one month. The perspective is to concomitantly evaluate technical and non-technical performance, and the impact of stress on both. This is the first randomized trial studying repetition of simulation sessions and its impact on both clinical performance and stress as explored by objective and subjective assessments. The investigators expect that stress decreases team performance and that repeated simulation increases team performance. The investigators expect no variation of stress parameters regardless of level of performance.

ELIGIBILITY:
Inclusion Criteria:

* Multidisciplinary team made up of 4 persons:

  1. an emergency physician with less than seven years of experience ,
  2. a resident,
  3. a nurse,
  4. and an ambulance driver.

Exclusion Criteria:

* Past history and/or psychiatric disease that modifies stress response,
* Pacemaker or implantable defibrillator,
* Treatment with a medication having a potential effect on stress parameters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Salivary Cortisol (SC) during high-fidelity simulation as measure of biological stress response | 1 year
Electrophysiological stress response profile made up of: Heart Rate (HR), Blood Pressure (BP), and Holter parameters (PNN50, HF/BH) during high-fidelity simulation | 1 year
Psychological stress response profile made up of: scores on State-Trait Anxiety Inventory (STAI), Impact of Event Scale - Revised (IES-R), Posttraumatic Stress Disorder Checklist Scale (PCLS) questionnaires during high-fidelity simulation | 1 year

SECONDARY OUTCOMES:
Effect of repetitive simulation sessions on technical skills performance profile made up of: scores of Team Average Performance Assessment Scale (TAPAS), IO access performance assessment scale | 1 year
Effect of repetitive simulation sessions on non-technical performance profile made up of: scores of Clinical Teamwork Scale (CTS), Behavioural Assessment Tool (BAT) | 1 year
Effect of repetitive simulation sessions on stress response profile made up of: SC, HR, BP, PNN50, HF/BH, STAI, IES-R, PCLS | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A GHAZALI, MD, Principal Investigator — University Hospital of Poitiers
Locations (1):
- GHAZALI, Poitiers, France

REFERENCES:
- [Derived] Ghazali DA, Breque C, Sosner P, Lesbordes M, Chavagnat JJ, Ragot S, Oriot D. Stress response in the daily lives of simulation repeaters. A randomized controlled trial assessing stress evolution over one year of repetitive immersive simulations. PLoS One. 2019 Jul 25;14(7):e0220111. doi: 10.1371/journal.pone.0220111. eCollection 2019. PMID 31344077
- [Derived] Ghazali DA, Darmian-Rafei I, Ragot S, Oriot D. Performance Under Stress Conditions During Multidisciplinary Team Immersive Pediatric Simulations. Pediatr Crit Care Med. 2018 Jun;19(6):e270-e278. doi: 10.1097/PCC.0000000000001473. PMID 29432402
- [Derived] Ghazali DA, Ragot S, Breque C, Guechi Y, Boureau-Voultoury A, Petitpas F, Oriot D. Randomized controlled trial of multidisciplinary team stress and performance in immersive simulation for management of infant in shock: study protocol. Scand J Trauma Resusc Emerg Med. 2016 Mar 25;24:36. doi: 10.1186/s13049-016-0229-0. PMID 27012938